CLINICAL TRIAL: NCT04930042
Title: A Randomized, Double-blind, Multicenter Study to Demonstrate Equivalent Efficacy and to Compare Safety and Immunogenicity of a Biosimilar Ustekinumab (AVT04) and Stelara® in Patients With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: Efficacy, Safety, and Immunogenicity of AVT04 With Moderate-to-Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVT04-GL-301
Record Dates: First submitted 2021-01-19; First posted 2021-06-18 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVT04 45 mg SC (Experimental): Test Product: AVT04 (ustekinumab) Initial loading dose of 45 mg followed by 45 mg SC once every 12 weeks starting 4 weeks after the initial loading dose administered SC. Injected as subcutaneous in thigh and abdomen.
  Interventions: Drug: AVT04
- EU Stelara 45 mg SC (Active Comparator): Comparator ref product: EU Stelara (ustekinumab) Initial loading dose of 45 mg followed by 45 mg SC once every 12 weeks starting 4 weeks after the initial loading dose administered SC. Injected as subcutaneous in thigh and abdomen.
  Interventions: Drug: Stelara

INTERVENTIONS:
Drug: Stelara — AVT04 or Stelara (45 mg/5ml) will be administered as a subcutaneous injection in the thigh or abdomen per the approved dosing regimen for moderate to severe chronic PsO for patients with a body weight ≤100 kg.11,12
  Arms: EU Stelara 45 mg SC
Drug: AVT04 — AVT04 or Stelara (45 mg/5ml) will be administered as a subcutaneous injection in the thigh or abdomen per the approved dosing regimen for moderate to severe chronic PsO for patients with a body weight ≤100 kg.11,12
  Arms: AVT04 45 mg SC

SUMMARY:
Safety and Efficacy study of AVT04 (Alvotech Biosimilar to Ustekinumab), in patients with moderate to severe plaque psoriasis

DETAILED DESCRIPTION:
AVT04 is a fully human immunoglobulin class G1κ monoclonal antibody that specifically binds to the shared p40 protein subunit of IL-12 and IL-23 and therefore inhibits their activites

AVT04 is being developed to be a biosimilar with the European Union (EU)-licensed drug Stelara® (hereafter referred to as Stelara) ustekinumab, Anatomical Therapeutic Chemical code: L04AC05) injection for subcutaneous (SC) and intravenous use. Stelara is an anti-IL-12 and anti-IL-23 monoclonal antibody approved for various indications. Indications approved in the EU11 and United States (US)12 include: PsO in adult and pediatric patients, psoriatic arthritis, Crohn's disease, and ulcerative colitis. Indications approved in the People's Republic of China include PsO and Crohn's disease.13 Approval status may differ in other geographic regions.

This is a multicenter, double-blind, randomized, active control clinical study to compare the efficacy, safety, and immunogenicity of AVT04 versus Stelara in patients with moderate to severe chronic PsO.

The active period of Study AVT04-GL-301 comprises 2 stages:

* Stage 1: Primary Efficacy Assessment (Day 1 to Week 15)
* Stage 2: Long Term Efficacy and Safety Assessment (Week 16 to 52) Stage 1 On Day 1, after successfully completing Screening activities, eligible patients will be randomized into Groups 1 and 2, in a 1:2 ratio (AVT04:Stelara), and begin Stage 1.

Patient randomization will be stratified by presence or absence of previous biologic treatment, by region; ie, Europe or China, and by body weight category (≤80 kg vs >80 kg).

* Group 1: Patients will receive an initial dose of AVT04 45 mg administered SC, followed by 45 mg 4 weeks later.
* Group 2: Patients will receive an initial loading dose of Stelara, 45 mg administered SC, followed by 45 mg 4 weeks later.

Stage 2

At Week 16:

Patients who were initially randomized in Group 1 (AVT04) will continue to receive AVT04 45 mg SC every 12 weeks at Weeks 16, 28, and 40 (unless withdrawn from the study).

Patients who were initially randomized in Group 2 (Stelara) will be re-randomized into Groups 2A and 2B, in a 1:1 ratio:

* Group 2A: Patients will begin receiving AVT04 45 mg SC every 12 weeks, at Weeks 16, 28, and 40 (unless withdrawn from the study).
* Group 2B: Patients will continue to receive Stelara 45 mg SC every 12 weeks, at Weeks 16, 28, and 40 (unless withdrawn from the study).

At Week 28:

* Non-responsive patients (PASI improvement <50% compared to BL) will be encouraged to continue in the study for safety analyses, per the Schedule of Assessments (SoA) (Table 7.1), but will not receive further study drug.
* Responsive patients (PASI improvement ≥50% compared to BL) will continue in the study.

At Week 40: All patients who are still in the study (except Week 28 non-responsive patients) will receive the final study drug administration.

At Week 52 (EoS/ET): All patients will undergo final efficacy and safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the informed consent form (ICF) and documentation as required by relevant competent authorities and is able to understand and adhere to the visit schedule and study requirements.
2. Chinese patients shall be recruited in Mainland China.
3. Patient is male or female, aged 18 to 75 years old, inclusive, at time of Screening.
4. Patient weighs ≤100 kg at Screening and at BL.
5. Patient has had moderate to severe chronic PsO for at least 6 months.
6. Patient has involved body surface area (BSA) ≥10%, PASI ≥12, and sPGA ≥3 (moderate) at Screening and at BL.
7. Patient has had stable psoriatic disease for at least 2 months (ie, without significant changes as defined by the investigator or designee) prior to Screening.
8. Patient is a candidate for systemic therapy because the patient has had a previous failure, inadequate response, intolerance, or contraindication to at least 1 systemic antipsoriatic therapy including, but not limited to, methotrexate, cyclosporine, psoralen plus ultraviolet light A (PUVA), and ultraviolet light B (UVB).
9. Patient has a negative QuantiFERON test for tuberculosis (TB) during Screening.

   Note: Patients with an indeterminate QuantiFERON test are allowed if they have all of the following:
   1. No evidence of active TB on chest radiograph within 3 months prior to the first dose of study drug.
   2. Documented history of adequate prophylaxis initiation prior to receiving study drug in accordance with local recommendations.
   3. No known exposure to active TB after most recent prophylaxis.
   4. Asymptomatic at Screening and BL. Investigators should check with the medical monitor before enrolling such patients.
10. Patient is naïve to ustekinumab therapy, approved or investigational.
11. Women of childbearing potential (except those who are postmenopausal for more than 2 years or if surgically sterile) must have a negative serum pregnancy test during Screening and negative urine pregnancy test at BL.

Sexually active women of childbearing potential must agree to use highly effective contraception (sterilization, hormonal contraception pills or injection or implants, and abstinence) for the duration of the study and until 4 months after the last dose of the study drug. Male patients must agree to use contraception for the duration of the study and agree not to donate sperm during and for 4 months after the last dose of study drug.

Note: Male partners of female subjects should also use contraception and should not donate sperm until 4 months after the last dose of study drug.

Exclusion Criteria:

1. Patient diagnosed with psoriatic arthritis, erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, other skin conditions (eg, eczema), or other systemic autoimmune disorder inflammatory disease at the time of the Screening Visit that would interfere with evaluations of the effect of the study drug on psoriasis.
2. Patient has prior use of any of the following medications within specified time periods or will require use during the study:

   1. Topical medications within 2 weeks of BL visit (except low- to mid-potency topical corticosteroids on face, eyes, scalp, palms, soles, and genital area; only).
   2. PUVA phototherapy and/or UVB phototherapy within 4 weeks prior to the BL visit.
   3. Nonbiologic psoriasis systemic therapies (eg, cyclosporine, methotrexate, and acitretin) within 4 weeks prior to the BL visit.
   4. Any systemic steroid in the 4 weeks prior to the BL visit.
   5. Any oral traditional Chinese medicine (TCM) 4 weeks prior to the BL visit or any topical TCM 2 weeks prior to the BL visit.
   6. Investigational agent(s) within 90 days or 5 half-lives (whichever is longer) before BL visit.
   7. Other systemic biologics within 90 days or 5 half-lives (whichever is the longer) before BL visit.
   8. Any therapeutic agent targeting IL-12, IL-17 or IL-23 at any time. Specified washout periods for approved/marketed products are provided in Table 5.1.

   Table 5.1: Approved/Marketed Products Medication or Therapy Washout before BL Biologic Therapies, including but limited to: Adalimumab Etanercept Secukinumab Infliximab Certolizumab pegol Alefacept Briakinumab Guselkumab Brodalumab 12 weeks 8 weeks 12 weeks 12 weeks 24 weeks 24 weeks 24 weeks 13 weeks 13 weeks Any kinase inhibitor for any reason (eg, tofacitinib citrate) 1 day Any phosphodiesterase type 4 inhibitor (eg, apremilast [Otezla]) 4 weeks Cyclosporine 4 weeks Methotrexate 4 weeks PUVA-UVA/UVB 4 weeks Topical psoriasis treatments (examples include vitamin D analogs, topical steroids, polifenols, etc) (except low- to mid-potency topical corticosteroids on face, eyes, scalp, palms, soles, and genital area; only) 2 weeks Oral retinoids 4 weeks Corticosteroids IM - IV - oral - intraarticular 4 weeks Drugs that may cause new onset or exacerbation of psoriasis (including, but not limited to, beta blockers, lithium, and anti-malarials) 6 months1 TCM (oral) TCM (topical) 4 weeks 2 weeks Abbreviations: BL = Baseline; IM = intramuscular; IV = intravenous; PUVA = psoralen plus ultraviolet light A; TCM = traditional Chinese medicine; UVA = ultraviolet light A; UVB = ultraviolet light B. 1 Unless the patient has been on a stable dose for at least 6 months prior to BL Visit without exacerbation of psoriasis.
3. Patient has received live or attenuated vaccines during the 4 weeks prior to BL visit or has the intention of receiving a live or attenuated vaccine at any time during the study.

   Note: Inactivated (non-live and non-attenuated) vaccines are allowed.
4. Patient has an underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious, or gastrointestinal) which, in the opinion of the investigator or designee, significantly immunocompromises the patient and/or places the patient at unacceptable risk for receiving an immunomodulatory therapy.
5. Patient has a planned surgical intervention during the duration of the study except those related to the underlying disease and which, in the opinion of the investigator or designee, will not put the patient at further risk or hinder the patient's ability to maintain compliance with study drug and the visit schedule.
6. Patient has an active and serious infection or history of infections as follows:

   a. Any active infection (including Severe Acute Respiratory Syndrome-Coronavirus-2 [SARS-CoV-2] infection) i. For which non-systemic anti-infectives were used within 4 weeks prior to BL visit. Note: patients receiving topical antibiotics for facial acne do not need to be excluded.

   ii. Which required hospitalization/quarantine or systemic anti-infective within 8 weeks prior to BL visit.

   b. Recurrent or chronic infections or other active infection that, in the opinion of the investigator or designee, might cause this study to be detrimental to the patient.

   c. Invasive fungal infection or mycobacterial infection. d. Opportunistic infections, such as listeriosis, legionellosis, or pneumocystis.
7. Patient is positive for human immunodeficiency virus (HIV), hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb).
8. Patient has severe progressive or uncontrolled, clinically significant disease that in the judgment of the investigator or designee renders the patient unsuitable for the study.
9. Patient has a history of malignancy within 5 years except for adequately treated cutaneous squamous or basal cell carcinoma, in situ cervical cancer or in situ breast ductal carcinoma.
10. Patient has active neurological disease such as multiple sclerosis, Guillain-Barré syndrome, optic neuritis, transverse myelitis, or history of neurologic symptoms suggestive of central nervous system demyelinating disease.
11. Patient has moderate to severe heart failure (New York Heart Association class III/IV).
12. Patient has uncontrolled diabetes mellitus type 1 or 2.
13. Patient has a history of hypersensitivity to the active substance or to any of the excipients of Stelara or AVT04.
14. Patient is pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation.
15. Patient has evidence (as assessed by the investigator or designee using good clinical judgment) of alcohol or drug abuse or dependency at the time of Screening, for the 5 years prior to Screening, or during the study.
16. Patient is unable to follow study instructions and comply with the protocol in the opinion of the investigator or designee.
17. Patient has a history of clinically significant hematological abnormalities, including cytopenia (eg, thrombocytopenia, leukopenia).
18. Patient has a laboratory abnormality that, in the opinion of the investigator or designee, could cause this study to be detrimental to the patient. The following laboratory abnormalities should be excluded:

    1. Hemoglobin <9 g/dL
    2. Platelet count <100,000/mm³
    3. White blood cell count <3000 cells/mm³
    4. Aspartate aminotransferase and/or alanine aminotransferase that is persistently ≥2 × the upper limit of normal. (Persistently indicates at least on 2 occasions separated by a number of days, per the rescreening procedure)
    5. Creatinine clearance <50 mL/min (Cockcroft-Gault formula)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Baseline to week 12
  Percent (%) change in Psoriasis Area and Severity Index (PASI)

SECONDARY OUTCOMES:
PASI 50, 75, 90 and 100 response rates | Baseline to week 52
  PASI 50, 75, 90, and 100 response rates at Weeks 4, 8, 12, 16, 28, 40, and 52 (EoS/ET)
PASI percent improvement | Baseline to week 52
  Percent improvement in PASI from BL to Week 4, 8, 16, 28, 40, and 52 (EoS/ET).

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldmann, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (30):
- Estonia (3):
  - North Estonia Medical Centre, Tallinn
  - Innomedica OU, Tallinn
  - Tartu University Hospital, Tartu
- Georgia (6):
  - Aleksandre Aladashvili Clinic, LLC, Tbilisi
  - J.S.C. Curatio, Tbilisi
  - LEPL The First University Clinic of Tbilisi State Medical University, Tbilisi
  - Scientific Research National Center of Dermatology and Venereology LLC, Tbilisi
  - Health Institute LLC, Tbilisi
  - David Abuladze Georgian-Italian Clinic LTD, Tbilisi
- Poland (14):
  - ClinicMed Daniluk, Nowak Spolka Jawna, Bialystok
  - Centrum Badan Klinicznych PI-House Sp. Z o.o, Gdansk
  - Centrum Medyczna ALL-MED, Krakow
  - SGD SC, Krakow
  - DERMED Centrum Medyczne Sp. z o.o., Lodz
  - Dermoklinika Centrum Medyczne s.c. M.Kierstan, J. Narbutt, A. Lesiak, Lodz
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Kliniczny Szpital Wojewódzki Nr. 1 im. Fryderyka Chopina, Klinika Detmatologii, Rzeszów
  - MICS Centrum Medyczne Toruń, Torun
  - Medycyna Kliniczna, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - DermMedica Sp. z o.o, Wroclaw
  - WroMedica I. Bielicka, A. Strzalkowska s.c., Wroclaw
- Ukraine (7):
  - Communal nonprofit enterprise ,,City Dermatovenereological Dispensary #2,, Kharkiv city council, Kharkiv
  - Private Medical Center Medical Clinic Blagomed LLC, Kyiv
  - National Medical University named after O.O.Bohomolets, Kyiv
  - Treatment and Diagnostic Center of private enterprise "Asclepius", Lviv
  - Municipal Enterprise "Rivne Regional Dermatology and Venereology Dispensary" of Rivne Regional Council, Rivne
  - Treatment and Diagnostic Center of private enterprise "Asclepius", Uzhhorod
  - Military Hospital (Military Unit A3309) of Military-Medical Clinical Center of Eastern Region, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feldman SR, Reznichenko N, Berti F, Duijzings P, Ruffieux R, Otto H, Haliduola HN, Leutz S, Stroissnig H. Randomized, double-blind, multicenter study to evaluate efficacy, safety, tolerability, and immunogenicity between AVT04 and the reference product ustekinumab in patients with moderate-to-severe chronic plaque psoriasis. Expert Opin Biol Ther. 2023 Jul-Dec;23(8):759-771. doi: 10.1080/14712598.2023.2235263. Epub 2023 Jul 12. PMID 37435850